CLINICAL TRIAL: NCT02051439
Title: A Comparison of the Party Balloon Assisted Valsalva With Conventional Valsalva Maneuver in Diagnosis of Superficial Venous Valvular Reflux of Lower Limb
Brief Title: The Party Balloon Assisted Valsalva in Diagnosis of Superficial Venous Valvular Reflux of Lower Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SIRIRAJ11SU00030/028/11
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Varicose Veins; Venous Insufficiency
Keywords: Varicose Veins; Venous Insufficiency; Doppler; Duplex; Valsava
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valsava (Other): The patients were randomized to 2 groups. The first group performed conventional Valsava before balloon assisted Valsava. The second group performed balloon assisted Valsava before conventional Valsava for venous reflux examination by duplex scan.
  Interventions: Procedure: Valsava

INTERVENTIONS:
Procedure: Valsava — The patients were randomized to 2 groups. The first group performed conventional Valsava 3 times before balloon assisted Valsava 3 times. The second group performed balloon assisted Valsava 3 times before conventional Valsava 3 times for venous reflux examination by duplex scan.

SUMMARY:
This study was designed to compare the party balloon assisted Valsalva with the conventional Valsava for exhibiting the reverse venous flow in superficial venous valvular incompetence duplex examination.

DETAILED DESCRIPTION:
In this study, we compared the Party Balloon assisted Valsalva with Conventional Valsalva maneuver in diagnosis of superficial venous valvular reflux of lower limb by crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Age within 18-80 years old
* Visible GSV varicose veins
* Trendelenburg test part 1 - Negative (Perforator vein incompetence) and
* Trendelenburg test part 2 - Positive (Saphenofemoral junction competence)
* Consent to participate in the study.

Exclusion Criteria:

* - CVI from Klippel-Trenaunay syndrome, Deep vein thrombosis (DVT), Arteriovenous fistula (AVF)
* Failure to language communication
* Previous heart disease (CAD, Myocardial infarction, Stable angina, Unstable angina, Congestive Heart Failure, Valvular heart disease)
* Previous lung disease (Asthma, Chronic obstructive pulmonary disease, Bronchiectasia)
* Abnormalities of oral cavity which cannot hold own breath. (Cleft lip, Cleft palate)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of successfully identified reflux with different method of Valsava technic | 20 minutes
  Patients performed conventional Valsava for identify venous reflux on duplex scan for 3 times then they performed balloon assisted Valsava for identify venous reflux on duplex scan for 3 times. The Outcome is number of successfully identified reflux with different method of Valsava technic.

SECONDARY OUTCOMES:
The timing for the instruction of conventional Valsava and balloon assisted Valsava | 20 minutes
  The time for training patients to performed conventional Valsava and balloon assisted Valsava before duplex examination was compared
The timing of identified venous reflux demonstrated in the duplex scan of conventional Valsava and balloon assisted Valsava | 20 minutes
  The time of identified venous reflux demonstrated in the duplex scan of conventional Valsava and balloon assisted Valsava was compared
The total timing for duplex scan examination in conventional Valsava and balloon assisted Valsava | 20 minutes
  The total timing for duplex scan examination in conventional Valsava and balloon assisted Valsava was compared